CLINICAL TRIAL: NCT00691353
Title: Subjective Well Being of Patients Receiving Atypical Antipsychotics as Monotherapy or Cotherapy With Mood Stabilizers
Acronym: DIDAXI
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Pontikis Panagiotis, MD Medical and Regulatory Affairs Director, AstraZeneca, SA Greece
Other Study IDs: NIS-NGR-DUM-2008/1
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-12

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; antipsychotics; social functioning; mood stabilizers; Bipolar Disorder Type I; atypical antipsychotics; monotherapy; cotherapy
MeSH Terms: conditions — Bipolar Disorder; Social Adjustment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Cross - Sectional study requiring one visit at the investigators office for the data collection.

* Target Group: Patients that suffer from Bipolar Disorder Type 1.
* YMRS - HAMILTON and GAF scales are going to be used to assess the clinical outcome. The findings are going to be based on the different scores reported by Specialists (before the patients started to use as a therapy atypical antipsychotics / at the time that the visit actually takes place for the cause of the study.) We predefine the time period that the patient should be using atypical antipsychotics at minimum (2 months).
* The first 9 consecutive patients that visit the Specialist and meet the entry criteria and signs the ICF will be recruited in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are diagnosed with Bipolar Disorder Type 1 according to diagnostic criteria DSM - IV
* Patients that have started therapy with atypical antipsychotics as monotherapy or cotherapy with mood stabilizers the last three months, but have completed 2 full months of therapy.
* Patients with anxiety disorder can be recruited in the study unless it is dominant.

Exclusion Criteria:

* Patients that use antidepressant medication
* Patients who were treated with depot antipsychotic in the last quarter before their enrollment in the study.
* Patients who are addicts of toxic substances.
* Patients who suffer from other serious diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target Group:Patients that suffer from Bipolar Disorder Type 1 who are treated with atypical antipsychotics as monotherapy or cotherapy with mood stabilizers
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Difference in the scores reported in YMRS and Hamilton - D scales from baseline(start of therapy) | Assessment of the progress of disease 2 to 4 months after the initiation of the therapy(baseline)
Assessment of functioning - Relative score reported in GAF scale | 2 - 4 months after the initiation of the therapy. No baseline comparison

SECONDARY OUTCOMES:
To depict sociodemographic characteristics and comorbidities. | Reported at the site visit

CONTACTS AND LOCATIONS:
Overall Officials: Charalambos Touloumis, MD, Principal Investigator — Athens Psychiatric Hospital Greece
Locations (20):
- Greece (20):
  - Research Site, Agrinio
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Crete
  - Research Site, Elefsina
  - Research Site, Ioannina
  - Research Site, Karditsa
  - Research Site, Katerini
  - Research Site, Kos
  - Research Site, Kozani
  - Research Site, Lamia
  - Research Site, Larissa
  - Research Site, Nafplion
  - Research Site, Pátrai
  - Research Site, Piraeus
  - Research Site, Rhodes
  - Research Site, Serres
  - Research Site, Thebes
  - Research Site, Thessalonii
  - Research Site, Thessaloniki